CLINICAL TRIAL: NCT05076357
Title: Cold Exposure, Appetite Control and Weight Loss in Individuals Living With Obesity
Brief Title: Cold, Appetite and Weight Loss in Individuals With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Eric Doucet, Full Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-09-19-4928
Record Dates: First submitted 2021-04-26; First posted 2021-10-13 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Weight Loss; Cold Exposure; Appetitive Behavior
Keywords: weight loss; appetite; cold exposure; obesity; nutritional intervention
MeSH Terms: conditions — Weight Loss; Appetitive Behavior; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: This study is an 8 week weight loss intervention with 3 randomly assigned groups: DIET, cold exposure (CE), and DIET+CE. Participants in the CE and DIET+CE groups will report to the laboratory every 2nd day for the 8 week intervention to undergo cold exposure. The DIET and DIET+CE groups will have a weekly nutritional consultation at the lab as well as a weekly check-in with the nutritionist via text, phone, or email.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only diet group (Experimental): Dietary energy prescription at -30% of Energy requirements (50% carbohydrate; 30% fat; 20% protein) during 8 weeks. Follow up with a registered dietitian.
  Interventions: Behavioral: Caloric Restriction
- Only cold exposure group (Experimental): No dietary intervention. Visit at laboratory every 2nd day during the 8-week intervention to undergo the cold exposure as follows: 2 weeks of exposure at 18 degrees, 2 weeks of exposure at 14 degrees and 4 weeks of 10 degrees of exposure during 90 min.
  Interventions: Other: Cold intervention
- Combined diet + cold exposure group (Experimental): Dietary energy prescription at -30% of Energy requirements (50% carbohydrate; 30% fat; 20% protein). Follow up with a registered dietitian. Visit at laboratory every 2nd day during the 8-week intervention to undergo the cold exposure as follows: 2 weeks of exposure at 18 degrees, 2 weeks of exposure at 14 degrees and 4 weeks of 10 degrees of exposure during during 90 min.
  Interventions: Behavioral: Caloric Restriction

INTERVENTIONS:
Behavioral: Caloric Restriction — -30% of participants total energy requirements
  Arms: Combined diet + cold exposure group; Only diet group
Other: Cold intervention — Sessions of 90min each every 2nd day involving cold exposure
  Arms: Only cold exposure group

SUMMARY:
This study is an 8 week weight loss intervention with 3 randomly assigned groups: DIET, cold exposure (CE), and DIET+CE. The study will be a total of 13 weeks. All participants will undergo a screening session, two experimental sessions at baseline and two experimental sessions after the intervention.

There will be a control (ambient) experimental session and a cold exposure experimental session These will be done in a randomized order both before and after the intervention. Therefore, a total of 5 lab visits will be required for all participants regardless of group outside of their assigned group intervention. Participants in the CE and DIET+CE groups will report to the laboratory every 2nd day for the 8 week intervention to undergo cold exposure as outlined below. The DIET and DIET+CE groups will have a weekly nutritional consultation at the lab as well as a weekly check-in with the nutritionist via text, phone, or email. Participants will be randomly assigned a group after completing the screening session and prior to the experimental session.

DETAILED DESCRIPTION:
This study is an 8 week weight loss intervention with 3 randomly assigned groups: DIET, cold exposure (CE), and DIET+CE. The study will be a total of 13 weeks. All participants will undergo a screening session outlined below. There will be 4 experimental sessions, 2 before and 2 after the intervention. There will be one week between each session. The timeline will be:

* Screening
* Experimental session 1
* Experimental session 2
* Intervention
* Experimental session 3
* Experimental session 4. There will be a control (ambient) experimental session and a cold exposure experimental session (outlined below). These will be done in a randomized order both before and after the intervention. Therefore, a total of 5 lab visits will be required for all participants regardless of group outside of their assigned group intervention. Participants in the CE and DIET+CE groups will report to the laboratory every 2nd day for the 8 week intervention to undergo cold exposure as outlined below. The DIET and DIET+CE groups will have a weekly nutritional consultation at the lab as well as a weekly check-in with the nutritionist via text, phone, or email. Participants will be randomly assigned a group after completing the screening session and prior to the experimental session. Participants cannot be assigned prior to consenting, as this will bias the randomization process and make it irrelevant. They will have all 3 groups explained to them prior to consenting but will not be assigned until after screening.

SCREENING Informed consent will be collected and verification of inclusion criteria. Participants will be invited to rate the food items the most consume from different categories: high fat sweet, low fat sweet, high fat savory, low fat savory. The results will be used for the Leeds Food preference Questionnaire (LFPQ) that will be applied in the experimental sessions. Measures of height and weight will be collected. Afterwards, participants will be given an accelerometer (Actical-Mini Mitter Co. Inc.) to measure their activity levels for 1 week.

EXPERIMENTAL SESSIONS 7h15 - Anthropometrics and DEXA. Participants will be asked to arrive after a 12h overnight fast and having refrained from vigorous activities for 48h. Body weight and height (HR-100 Height Rod and BWB-800AS Digital Scale, Tanita Corporation of America, Inc. Arlington Heights, Illinois, USA) will be measured. A Dual Energy X-Ray Absorptiometry (DEXA) (Lunar Prodigy, GE Medical Systems).scan will be used to measure bone density, fat mass and lean body mass. Participants will have to lie on an examination table, fully clothed, while a low intensity x-ray will scan the entire body. The measurements take 15 minutes.

7h30 - Insertion of catheter. A qualified nurse will place an intravenous catheter into the ante-cubital vein distal to the elbow to take blood draws at various points outlined below. A total of X collections will be done, with each collections being 10 mL for a total of 80 mL. The first will be taken immediately after insertion. This will be followed by a short rest period. Blood samples will be kept for 10 years after publication, and then will be destroyed through the university biohazard waste disposal process. Blood draws will occur at the following additional time points: 9h, 9h40, 10h20, 11h, 11h40, 12h20, 1h..

8h00 - Resting energy expenditure. Participants will be asked to undergo a shortened version of the resting energy expenditure measurement outlined above, lasting approximately 30 minutes.

8h30 - Appetite measurement. Participants will be asked to fill out visual analog scales (VAS) at this point and various other points during the session. Briefly, desire to eat, hunger, fullness and prospective food consumption will be rated. Questions will be asked as follows: 1) "How strong is your desire to eat?" (Very weak- Very strong); 2) "How hungry do you feel?" (Not hungry at all- As hungry as I have ever felt); 3) "How full do you feel?" (Not full at all- Very full), and 4) "How much food do you think you could eat?" (Nothing at all- A large amount). VAS will be completed at the following additional time points: 9h, 9h40, 10h20, 11h, 11h40, 12h20, 1h.

8h35 -Participants will be served a standard breakfast including two pieces of toasts, jam, peanut butter, orange juice . They will be served the same breakfast for each session. They must consume the entirety of its contents within 20 minutes.

9h00 - Baseline measurements. Participants will be fitted with 4 surface electrodes (Delsys, Boston, MA, 02215, USA) on their sternocleidomastoid, trapezius, pectoralis major, and rectus abdominis to measure muscular activity during shivering. They will do 3 maximal contractions of 5 seconds for each muscle to create a baseline measurement for comparison. They will then be fitted with 12 thermocouples (Concept Engineering, Old Saybrook, CT) at the following sites: forehead, upper back, lower back, abdominal area, quadriceps, hamstrings, front calf, back calf, chest, biceps, forearm, and hand. These thermocouples measure skin temperature and get an overall mean skin temperature (Tskin). They will then be fitted with a 3 piece liquid conditioned suit (LCS: Three Piece, Allen Vangard, Ottawa, ON, Canada) that can be infused with either cold or ambient temperature water to manipulate skin temperature. Tskin will be measured at rest while participants lay down on a bed to determine ambient Tskin. During this time the plexiglass hood will be placed over their head to measure energy expenditure. During this measurement, participants will lie still on their back with a plexiglass hood over their head in a quiet room using a flow controller and gas analyzer (FlowKit-500, FMS, Sable System International, Las Vegas, NV, USA). The expired air will be sampled to determine oxygen consumption and resting energy expenditure will be derived. This test requires that participants lie quietly and relaxed for approximately 60 minutes. They will also be asked to rate both thermal comfort and thermal sensation on scales of - to +5 during the exposure.

10h00 - Exposure. Participants will then undergo either CE or AC. For CE, the suit will be perfused with cold water (at 10°C) for 2h. For AC, the suit will be perfused with thermoneutral (33°C) water to maintain Tskin. During this, Tskin will be continually monitored, thermal comfort (i.e. how comfortable or uncomfortable you feel) and thermal sensation (i.e. how warm or cold you feel) will be measured every 5 minutes. We have previously shown that lean individuals in the suit with water at 5°C have no change in core temperature (i.e. compensable CE), meaning although participants were cold and uncomfortable, they were at no risk for freezing or non-freezing cold injuries. These general occur at a Tskin below 15°C, whereas a study we conducted using 5°C water in the suit achieved a lowest skin temperature of 24°C. The cold stimuli being used will make participants mildly uncomfortable but pose minimal risk of adverse events, although extreme evens that occur below the 15°C Tskin were listed for transparency. Participants are free to end the session if necessary, and there are blankets and hot shower facilities should they be needed. Once the exposure is completed, the suit, electrodes and thermocouples will all be removed.

13h00 - Olfaction and food reward. Participants will be required to complete 3 different odor tests using Sniffin' Sticks (Burghart Instruments, Wedel, Germany). This will test for odor identification, detection threshold, and discrimination. It has been shown that these tests are correlated with changes in food intake during weight loss, showing changes in the desirability of food. For the food reward task, participants will do the Leeds Food Preference Questionnaire. This is a computerized task that uses 16 foods in 4 different categories: high-fat sweet, low-fat sweet, high-fat non-sweet, low-fat non-sweet. Explicit values will be determined using a visual analog scale of 0-100, while implicit values will be determined by having the participant choose a preferred of 2 options on repeat, until all 16 foods have been matched with each other food. This allows for preference fat and sweet content of food to be compared.

13h30 - Ad Libitum lunch. Participants will be given a food menu, from which they can choose as many foods as they would like. They will all be served in ad libitum quantities, where they can consume as much or as little of each food as they would like in the given time period.

14h15 - Olfaction and food reward. The tasks listed above will be administered again.

14h45 - Conclusion. At the end of the trial participants will be asked to select foods to consume for the following two days from the validated food menu. They will be packed into labeled lunch boxes (coolers) and provided in ad libitum quantities, meaning they can consume as much or as little of each food as they would like, leaving any extra food, scraps, and wrappers in the cooler. Ad libitum food will be provided at the conclusion of each of the 4 experimental sessions. Food is not provided during the intervention.

DIET Intervention A 30% dietary restriction will be determined using the participant's resting energy expenditure (REE), accelerometer data (PA) and a coefficient of 1.10 for the thermic effect of feeding to calculate the energy required to maintain current body weight. This will be multiplied by a coefficient of 0.70. The formula will be: ((REE+PA)*1.10)*0.70. The diet will be prescribed by a nutritionist using the Canadian Food Exchange System. This will allow participants to select foods they enjoy during the weight loss, however in smaller quantities. Exchange lists are groups of foods that contain a similar mix of carbohydrates, protein, fat, and calories. The Canadian exchange system there are seven exchange groups: Grains & Starches; Fruits; Milk & Alternatives; Vegetables; Meat & Alternatives; Fats; Unlimited consumption. Within any group, you can exchange one food serving for another. The number of portions from each group will be recommended based on the macronutrient composition evaluated in the preliminary session. This session will also be used to clarify any potential questions regarding the project and the intervention. There will also be weekly sessions with the nutritionist of roughly 30 minutes at the lab, as well as mid-week check-in via text, email, or phone call to ensure compliance and provide support with the nutritionist.

COLD EXPOSURE Intervention Participants will come to the laboratory every second day during the 8 week intervention for a 90 minute session in the liquid conditioned suit, where the suit will be perfused with 10°C water. Again, this will be a compensable cold stimulus meaning there are no changes to core temperature. Participants will be free to move and talk during the intervention as EE is not being measured, although they will be either sitting or lying down during each session. They will be allowed to bring their own entertainment and Netflix will be provided. At the conclusion of the study there will be a consultation session with the nutritionist to explain the Canadian Food Exchange System, as well as answer dietary questions to provide balance with the DIET groups.

DIET+CE Intervention Participants will undergo both the dietary restriction of the diet group and the cold intervention of the CE group, described above.

ELIGIBILITY:
Inclusion Criteria:

* Present a 27≥BMI,
* Present a waist circumference >88 cm
* Must be weight-stable (±2 kg last 6 months)
* Must be sedentary (<2 times/week of 30 min of continuous exercise)
* Must be able to read in English
* Must to present no history of alcohol or drugs abuse

In addition, Women will be included if:

• Must be pre-menopausal with a regular menstrual cycle

Exclusion Criteria:

* present any history or evidence of cardiovascular disease
* present any history or evidence of peripheral vascular disease
* present any history or evidence of stroke
* present a current diagnosis of an axis 1 psychiatric disorder (i.e. mood, anxiety and eating disorders);
* be insulin dependent (75g oral glucose tolerance test)
* present a known renal and/or liver disease
* asthma requiring therapy
* plasma cholesterol > 8 mmol/L
* systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg
* present previous history of inflammation disease
* present previous history of cancer
* present untreated thyroid or pituitary disease
* present a regular consumption of medications that could affect cardiovascular function and/or metabolism (i.e. MAO inhibitors, pressor agents, warfarin, anticonvulsants, phenylbutazone, or tricyclic antidepressants)
* present food allergies
* be smoker
* present alcohol intake that exceeds recommendations or alcoholism
* present current addictions to opiates, cocaine or stimulants
* be pregnant or planning to become pregnant over the course of the study
* be peri- or post-menopausal
* have had surgically induced menopause

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline energy intake at 8 weeks | 8 weeks
  Energy intake will be measured both in the laboratory and in the free-living state for 3 days with a validated food menu (McNeil, 2012) and the Food Processor SQL from ESHA Research, Inc. Measures will be taken at baseline and after intervention.
Change from baseline in fasting hunger using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of fasting hunger using Visual Analogue scales will be performed in fasting state (12h) at baseline and in the end of the weight loss intervention
Change from baseline in fasting desire to eat using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of fasting desire to eat using Visual Analogue scales will be performed in fasting state (12h) at baseline and in the end of the weight loss intervention
Change from baseline fasting fullness using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of fasting fullness using Visual Analogue scales will be performed in fasting state (12h) at baseline and in the end of the weight loss intervention
Change from baseline in fasting prospective food consumption using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of fasting prospective food consumption using Visual Analogue scales will be performed in fasting state (12h) at baseline and in the end of the weight loss intervention
Change from baseline in post-prandial hunger using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of post-prandial hunger using Visual Analogue scales will be taken at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention
Change from baseline in post-prandial desire to eat using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of post-prandial desire to eat using Visual Analogue scales will be taken at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention
Change from baseline in post-prandial fullness using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of post-prandial fullness using Visual Analogue scales will be taken at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention
Change from baseline in post-prandial prospective food consumption using Visual Analogue scales at 8 weeks | 8 weeks
  Measures of post-prandial prospective food consumption using Visual Analogue scales will be taken at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention

SECONDARY OUTCOMES:
Change from baseline in Resting energy expenditure at 8 weeks | 8 weeks
  Resting energy expenditure will be measured at baseline and in the end the intervention
Changes from baseline in post-prandial explicit liking using the LFPQ at 8 weeks | 8 weeks
  explicit liking will be measured using a tool called Leeds Preference Food Questionnaire. Measures will be taken at baseline and at the end of the intervention
Changes from baseline in post-prandial explicit wanting using the LFPQ at 8 weeks | 8 weeks
  explicit wanting will be measured using a tool called Leeds Preference Food Questionnaire. Measures will be taken at baseline and at the end of the intervention
Changes from baseline in post-prandial implicit wanting using the LFPQ at 8 weeks | 8 weeks
  implicit wanting will be measured using a tool called Leeds Preference Food Questionnaire. Measures will be taken at baseline and at the end of the intervention
Changes from baseline in olfaction using the 'Sniffin Sticks' tests at 8 weeks | 8 weeks
  Olfaction will be measured using the Sniffin' Sticks (Burghart Instruments, Wedel, Germany), a 3-test battery of odorized markers that measure odor detection threshold, odor discrimination, and odor identification at 90 min after breakfast at baseline and after intervention
Changes from baseline in shivering response activity at 8 weeks | 8 weeks
  Changes in shivering response will be measured by surface electromyography (Delsys, Boston, MA, 02215, USA) from 7 muscles on the right side of the body:
  trapezius, latissimus dorsi, pectoralis major, vastus lateralis, rectus femoris, vastus medialis, and biceps femoris. EMG will be collected at 1000Hz and analyzed using a custom-designed MATLAB algorithms (Mathworks, Natick, MA) at baseline and after intervention.
Changes from baseline in thermal comfort at 8 weeks | 8 weeks
  Changes in thermal comfort will be measured using a LIKERT scale type (-5 to +5) at baseline and after the intervention
Changes from baseline in thermal sensation at 8 weeks | 8 weeks
  Changes in thermal sensation will be measured using a LIKERT scale type (-5 to +5) at baseline and after the intervention
Changes from baseline in total Ghrelin (EZGRT-89K) at 8 weeks | 8 weeks
  Blood samples will be collected fasting and at 30-min interval for 3 h in tubes containing EDTA and Aprotinin (anti-protease). Changes in total Ghrelin will be assayed with commercially available ELISA (Millipore, Billerica, MA 01821 USA) at baseline and after the intervention.
Changes from baseline in total Leptin (EZHL-80SK) at 8 weeks | 8 weeks
  Blood samples will be collected fasting and at 30-min interval for 3 h in tubes containing EDTA and Aprotinin (anti-protease). Changes in total Leptin will be assayed with commercially available ELISA (Millipore, Billerica, MA 01821 USA) at baseline and after the intervention.
Changes from baseline in total GLP-1 (EZGLP1T-36K) at 8 weeks | 8 weeks
  Blood samples will be collected fasting and at 30-min interval for 3 h in tubes containing EDTA and Aprotinin (anti-protease). Changes in total GLP-1 will be assayed with commercially available ELISA (Millipore, Billerica, MA 01821 USA) at baseline and after the intervention.
Changes from baseline in total PYY (EZHPYYT66K) at 8 weeks | 8 weeks
  Blood samples will be collected fasting and at 30-min interval for 3 h in tubes containing EDTA and Aprotinin (anti-protease). Changes in total PYY will be assayed with commercially available ELISA (Millipore, Billerica, MA 01821 USA) at baseline and after the intervention.
Changes from baseline in body composition at 8 weeks | 8 weeks
  Changes in body composition will be measured using a DXA (Lunar Prodigy, GE Medical Systems) at baseline and after intervention.
Changes from baseline in body weight at 8 weeks | 8 weeks
  Baseline and post intervention changes of body weight will be measured using a BWB-800AS Digital Scale from Tanita Corporation of America, Inc. Arlington Heights, Illinois, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Doucet, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No